CLINICAL TRIAL: NCT00025259
Title: A Phase III Groupwide Study of Dose-Intensive Response-Based Chemotherapy and Radiation Therapy for Children and Adolescents With Newly Diagnosed Intermediate Risk Hodgkin Disease
Brief Title: Chemotherapy With or Without Additional Chemotherapy and/or Radiation Therapy in Treating Children With Newly Diagnosed Hodgkin's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHOD0031; NCI-2011-02069 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000068943; COG-AHOD0031; AHOD0031 (Other: Childrens Oncology Group); AHOD0031 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2016-05

CONDITIONS: Childhood Lymphocyte-Depleted Classical Hodgkin Lymphoma; Childhood Mixed Cellularity Classical Hodgkin Lymphoma; Childhood Nodular Lymphocyte Predominant Hodgkin Lymphoma; Childhood Nodular Sclerosis Classical Hodgkin Lymphoma; Stage I Childhood Hodgkin Lymphoma; Stage II Childhood Hodgkin Lymphoma; Stage III Childhood Hodgkin Lymphoma; Stage IV Childhood Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Bleomycin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor; Prednisone; deltacortene; prednylidene; Vincristine

ARMS (7):
- Arm I (Patients off-therapy before callback-Induction only) (Experimental): Patients receive doxorubicin IV over 10-30 minutes on days 1-2, bleomycin sulfate IV over 10-20 minutes or SC and vincristine IV on days 1 and 8, etoposide IV over 1 hour on days 1-3, oral prednisone 2 or 3 times daily on days 1-7, and cyclophosphamide IV over 1 hour on day 1. Patients receive filgrastim (G-CSF) SC beginning on day 2 and continuing until blood counts recover (G-CSF is held on day 8). Treatment repeats every 21 days for 2 courses in the absence of progressive disease.
  Interventions: Biological: Bleomycin Sulfate; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Biological: Filgrastim; Drug: Prednisone; Drug: Vincristine Sulfate Liposome
- Arm II (RER with CR [ABVE-PC, IFRT]) (Experimental): Patients receive doxorubicin IV over 10-30 minutes on days 1-2, bleomycin IV over 10-20 minutes or SC and vincristine IV on days 1 and 8, etoposide IV over 1 hour on days 1-3, prednisone PO 2 or 3 times daily on days 1-7, and cyclophosphamide IV over 1 hour on day 1. Patients receive filgrastim (G-CSF) SC beginning on day 2 and continuing until blood counts recover (G-CSF is held on day 8). Treatment repeats every 21 days for 2 courses in the absence of progressive disease. Patients receive an additional 2 courses of ABVE-PC. Patients with sustained CR undergo IFRT approximately 3 weeks after the last day of ABVE course 4.
  Interventions: Biological: Bleomycin Sulfate; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Biological: Filgrastim; Radiation: Involved-Field Radiation Therapy; Drug: Prednisone; Drug: Vincristine Sulfate Liposome
- Arm III (RER with CR [ABVE-PC]) (Experimental): Patients receive doxorubicin IV over 10-30 minutes on days 1-2, bleomycin IV over 10-20 minutes or SC and vincristine IV on days 1 and 8, etoposide IV over 1 hour on days 1-3, prednisone PO 2 or 3 times daily on days 1-7, and cyclophosphamide IV over 1 hour on day 1. Patients receive filgrastim (G-CSF) SC beginning on day 2 and continuing until blood counts recover (G-CSF is held on day 8). Treatment repeats every 21 days for 2 courses in the absence of progressive disease. Patients receive an additional 2 courses of ABVE-PC. Patients with sustained CR are randomized to receive no further treatment.
  Interventions: Biological: Bleomycin Sulfate; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Biological: Filgrastim; Drug: Prednisone; Drug: Vincristine Sulfate Liposome
- Arm IV (RER with less than CR [ABVE-PC, IFRT]) (Experimental): Patients receive doxorubicin IV over 10-30 minutes on days 1-2, bleomycin IV over 10-20 minutes or SC and vincristine IV on days 1 and 8, etoposide IV over 1 hour on days 1-3, prednisone PO 2 or 3 times daily on days 1-7, and cyclophosphamide IV over 1 hour on day 1. Patients receive filgrastim (G-CSF) SC beginning on day 2 and continuing until blood counts recover (G-CSF is held on day 8). Treatment repeats every 21 days for 2 courses in the absence of progressive disease. Patients receive an additional 2 courses of ABVE-PC. Patients with VGPR, PR or SD undergo IFRT approximately 3 weeks after the last day of ABVE-PC course 4 for 5 days a week.
  Interventions: Biological: Bleomycin Sulfate; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Biological: Filgrastim; Radiation: Involved-Field Radiation Therapy; Drug: Prednisone; Drug: Vincristine Sulfate Liposome
- Arm V (RER with PD) (Experimental): Patients receive doxorubicin IV over 10-30 minutes on days 1-2, bleomycin IV over 10-20 minutes or SC and vincristine IV on days 1 and 8, etoposide IV over 1 hour on days 1-3, prednisone PO 2 or 3 times daily on days 1-7, and cyclophosphamide IV over 1 hour on day 1. Patients receive filgrastim (G-CSF) SC beginning on day 2 and continuing until blood counts recover (G-CSF is held on day 8). Treatment repeats every 21 days for 2 courses in the absence of progressive disease. Patients with PD are taken off therapy.
  Interventions: Biological: Bleomycin Sulfate; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Biological: Filgrastim; Drug: Prednisone; Drug: Vincristine Sulfate Liposome
- Arm VI (SER [DECA, ABVE-PC, IFRT]) (Experimental): Patients receive dexamethasone IV over 15 minutes, etoposide IV over 3 hours, and cytarabine IV over 3 hours on days 1-2. Patients receive 2 drops of dexamethasone ophthalmic solution every 6 hours on days 1, 2 and 3. Patients also receive cisplatin PO or IV over 12 hours as pre-hydration followed by continuous IV over 6 hours on day 1 and G-CSF SC beginning on day 3 and continuing until blood counts recover. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients then receive 2 additional courses of ABVE-PC chemotherapy. Patients with sustained complete or partial response undergo IFRT approximately 3 weeks after the last course of chemotherapy.
  Interventions: Biological: Bleomycin Sulfate; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Biological: Filgrastim; Radiation: Involved-Field Radiation Therapy; Drug: Prednisone; Drug: Vincristine Sulfate Liposome
- Arm VII (SER [ABVE-PC, IFRT]) (Experimental): Patients receive doxorubicin IV over 10-30 minutes on days 1-2, bleomycin IV over 10-20 minutes or SC and vincristine IV on days 1 and 8, etoposide IV over 1 hour on days 1-3, prednisone PO 2 or 3 times daily on days 1-7, and cyclophosphamide IV over 1 hour on day 1. Patients receive filgrastim (G-CSF) SC beginning on day 2 and continuing until blood counts recover (G-CSF is held on day 8). Treatment repeats every 21 days for 2 courses in the absence of progressive disease. Patients receive 2 additional courses of ABVE-PC. Patients with sustained complete or partial response undergo IFRT approximately 3 weeks after the last course of chemotherapy.
  Interventions: Biological: Bleomycin Sulfate; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Biological: Filgrastim; Radiation: Involved-Field Radiation Therapy; Drug: Prednisone; Drug: Vincristine Sulfate Liposome

INTERVENTIONS:
Biological: Bleomycin Sulfate — Given IV or SC
  Other Names: Blanoxan; BleMomycine; Blenoxane; Bleo-cell; Bleo-S; Bleocin; Bleolem; Bleomycin Sulfas; Bleomycin Sulphate; Blexane; Oil Bleo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm VI (SER [DECA, ABVE-PC, IFRT])
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: Arm VI (SER [DECA, ABVE-PC, IFRT])
Drug: Dexamethasone — Given IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
  Arms: Arm VI (SER [DECA, ABVE-PC, IFRT])
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Biological: Filgrastim — Given SC
  Other Names: Filgrastim XM02; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tbo-filgrastim; Tevagrastim
Radiation: Involved-Field Radiation Therapy — Undergo IFRT
  Other Names: IFRT; Involved field radiotherapy
  Arms: Arm II (RER with CR [ABVE-PC, IFRT]); Arm IV (RER with less than CR [ABVE-PC, IFRT]); Arm VI (SER [DECA, ABVE-PC, IFRT]); Arm VII (SER [ABVE-PC, IFRT])
Drug: Prednisone — Given orally
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone
Drug: Vincristine Sulfate Liposome — Given IV
  Other Names: Marqibo

SUMMARY:
This randomized phase III trial is studying different chemotherapy regimens given with or without radiation therapy to compare how well they work in treating children with newly diagnosed Hodgkin's disease. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Giving the drugs in different combinations may kill more cancer cells. Radiation therapy uses high-energy x-rays to damage cancer cells. It is not yet known if chemotherapy is more effective with or without additional chemotherapy and/or radiation therapy in treating Hodgkin's disease.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To compare response-based therapy to standard therapy for intermediate risk Hodgkin disease.

II. To determine whether involved field radiation therapy (IFRT) can be eliminated based upon early and complete response to multiagent chemotherapy.

III. To determine whether the addition of an additional two cycles of chemotherapy (DECA) can improve outcome in those with a slow early response to standard chemotherapy.

IV. To prospectively collect information on the individual prognostic significance of the following presenting factors: erythrocyte sedimentation rate, circulating levels of IL-10, each of the "B" symptoms - fever, night sweats, weight loss, nodal aggregate > 6 cm, large mediastinal mass > 1/3 thoracic diameter and number of involved nodal sites, histology, albumin, blood counts, sex and age.

V. To study the reliability and utility of [18F] -Fluorodeoxyglucose (FDG) Imaging (PET scans) as an imaging modality in Hodgkin disease.

VI. To determine the frequency and severity of late effects of therapy including thyroid dysfunction, infertility, cardiotoxicity, pulmonary toxicity and second malignant neoplasms.

VII. To serve as the therapeutic companion to biology studies in Hodgkin disease and correlate those results with response to therapy, event free-survival and overall survival.

OUTLINE: This is a randomized, multicenter study.

ARM I (ALL PATIENTS-OFF THERAPY BEFORE CALLBACK-INDUCTION CHEMOTHERAPY [ABVE-PC]): Patients receive doxorubicin intravenously (IV) over 10-30 minutes on days 1-2, bleomycin sulfate IV over 10-20 minutes or subcutaneously (SC) and vincristine IV on days 1 and 8, etoposide IV over 1 hour on days 1-3, oral prednisone 2 or 3 times daily on days 1-7, and cyclophosphamide IV over 1 hour on day 1. Patients receive filgrastim (G-CSF) SC beginning on day 2 and continuing until blood counts recover (G-CSF is held on day 8). Treatment repeats every 21 days for 2 courses in the absence of progressive disease. At the end of initial chemotherapy, patients undergo evaluation for response. Patients with less than 60% disease reduction are considered to have slow early response (SER). Patients with 60% or more disease reduction are considered to have rapid early response (RER).

RER: Patients receive 2 additional courses of ABVE-PC chemotherapy. After completion of treatment, patients are randomized to 1 of 4 treatment arms.

ARM II: Patients with sustained complete response (CR) undergo involved field radiation therapy (IFRT) approximately 3 weeks after the last day of ABVE-PC course 4 for 5 days a week.

ARM III: Patients with sustained CR receive no further treatment.

ARM IV: Patients with very good partial response (VGPR), partial response (PR) or stable disease (SD) undergo IFRT approximately 3 weeks after the last day of ABVE-PC course 4 for 5 days a week.

ARM V: Patients with progressive disease are taken off therapy and treated their physician's discretion.

SER: Patients are randomized to 1 of 2 treatment arms.

ARM VI: Patients receive dexamethasone IV over 15 minutes, etoposide IV over 3 hours, cytarabine IV over 3 hours on days 1-2, and receive 2 drops of dexamethasone ophthalmic solution every 6 hours on days 1, 2 and 3. Patients also receive cisplatin PO or IV over 12 hours as pre-hydration followed by continuous IV over 6 hours on day 1 and G-CSF SC beginning on day 3 and continuing until blood counts recover. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. After these 2 courses, patients then receive 2 additional courses of ABVE-PC chemotherapy.

ARM VII: Patients receive 2 courses of ABVE-PC chemotherapy.

In both SER arms, patients with sustained CR or PR undergo IFRT approximately 3 weeks after the last course of chemotherapy.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed, pathologically confirmed Hodgkin disease (all histologies) are eligible for this protocol if they meet the following clinical stage guidelines:

  * All Stage IB regardless of bulk disease
  * All Stage IIB regardless of bulk disease
  * Stage IA only with bulk disease
  * Stage IIA only with bulk disease
  * All Stage IAE, IIAE regardless of bulk disease
  * All Stage IIIA, IIIAE, IIIAS, IIIAE+S regardless of bulk disease
  * All Stage IVA, IVAE regardless of bulk disease
* May not be staged by laparotomy alone

  * Surgically staged patients must also have presurgical staging
* Bilirubin no greater than 1.5 times normal
* SGOT or SGPT less than 2.5 times normal
* Creatinine no greater than 1.5 times normal
* Creatinine clearance greater than 40 mL/min
* Radioisotope glomerular filtration rate greater than 70 mL/min
* Shortening fraction at least 27% by echocardiogram
* Ejection fraction at least 50% by MUGA
* No pathologic prolongation of QTc interval on 12-lead electrocardiogram
* FEV_1/FVC greater than 60% by pulmonary function test
* Pulse oximetry greater than 94%
* No evidence of dyspnea at rest
* No exercise intolerance
* Adequate venous access
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior chemotherapy
* At least 1 month since prior corticosteroids except prednisone for respiratory distress
* No prior radiotherapy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1734 (Actual)
Dates: Start 2002-09; Primary Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Friedman, Principal Investigator — Children's Oncology Group
Locations (175):
- United States (153):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - University of Florida, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Georgia Regents University Medical Center, Augusta, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health Richland, Columbia, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Science Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont College of Medicine, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Childrens Hospital-King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Clinic Children's Hospital, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (3):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (14):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - Chedoke Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Schneider Children's Medical Center of Israel, Petah Tikua, Israel
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- San Jorge Children's Hospital, San Juan, Puerto Rico
- Swiss Pediatric Oncology Group - Geneva, Geneva, Switzerland

REFERENCES:
- [Derived] Kreuzberger N, Goldkuhle M, von Tresckow B, Kobe C, Sickinger MT, Monsef I, Skoetz N. Positron emission tomography-adapted therapy for first-line treatment in adults with Hodgkin lymphoma. Cochrane Database Syst Rev. 2025 Mar 26;3(3):CD010533. doi: 10.1002/14651858.CD010533.pub3. PMID 40135712
- [Derived] Castellino SM, Giulino-Roth L, Harker-Murray P, Kahn JM, Forlenza C, Cho S, Hoppe B, Parsons SK, Kelly KM; COG Hodgkin Lymphoma Committee. Children's Oncology Group's 2023 blueprint for research: Hodgkin lymphoma. Pediatr Blood Cancer. 2023 Sep;70 Suppl 6(Suppl 6):e30580. doi: 10.1002/pbc.30580. Epub 2023 Jul 28. PMID 37505794
- [Derived] Johnston RL, Mottok A, Chan FC, Jiang A, Diepstra A, Visser L, Telenius A, Gascoyne RD, Friedman DL, Schwartz CL, Kelly KM, Scott DW, Horton TM, Steidl C. A gene expression-based model predicts outcome in children with intermediate-risk classical Hodgkin lymphoma. Blood. 2022 Feb 10;139(6):889-893. doi: 10.1182/blood.2021011941. PMID 34662378
- [Derived] Giulino-Roth L, Pei Q, Buxton A, Bush R, Wu Y, Wolden SL, Constine LS, Kelly KM, Schwartz CL, Friedman DL. Subsequent malignant neoplasms among children with Hodgkin lymphoma: a report from the Children's Oncology Group. Blood. 2021 Mar 18;137(11):1449-1456. doi: 10.1182/blood.2020007225. PMID 33512412
- [Derived] Welch JJG, Schwartz CL, Higman M, Chen L, Buxton A, Kanakry JA, Kahwash SB, Hutchison RE, Friedman DL, Ambinder RF. Epstein-Barr virus DNA in serum as an early prognostic marker in children and adolescents with Hodgkin lymphoma. Blood Adv. 2017 Apr 24;1(11):681-684. doi: 10.1182/bloodadvances.2016002618. eCollection 2017 Apr 25. PMID 29296710
- [Derived] Friedman DL, Chen L, Wolden S, Buxton A, McCarten K, FitzGerald TJ, Kessel S, De Alarcon PA, Chen AR, Kobrinsky N, Ehrlich P, Hutchison RE, Constine LS, Schwartz CL. Dose-intensive response-based chemotherapy and radiation therapy for children and adolescents with newly diagnosed intermediate-risk hodgkin lymphoma: a report from the Children's Oncology Group Study AHOD0031. J Clin Oncol. 2014 Nov 10;32(32):3651-8. doi: 10.1200/JCO.2013.52.5410. Epub 2014 Oct 13. PMID 25311218

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm VI (SER [DECA, ABVE-PC, IFRT]): Patients receive dexamethasone IV over 15 minutes, etoposide IV over 3 hours, & cytarabine IV over 3 hours on days 1-2. Patients receive 2 drops of dexamethasone ophthalmic solution every 6 hours on days 1, 2 & 3. Patients also receive cisplatin PO or IV over 12 hours as pre-hydration followed by continuous IV over 6 hours on day 1 & G-CSF SC beginning on day 3 & continuing until blood counts recover. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients then receive 2 additional courses of ABVE-PC chemotherapy. Patients with sustained complete or partial response undergo IFRT approximately 3 weeks after the last course of chemotherapy.
  Bleomycin Sulfate: Given IV or SC
  Cisplatin: Given IV
  Cyclophosphamide: Given IV
  Cytarabine: Given IV
  Dexamethasone: Given IV
  Doxorubicin Hydrochloride: Given IV
  Etoposide: Given IV
  Filgrastim: Given SC
  Involved-Field Radiation Therapy: Undergo IFRT
  Pre
Period: Overall Study
Arm/Group | Arm I (Patients Off-therapy Before Callback-Induction Only) | Arm II (RER With CR [ABVE-PC, IFRT]) | Arm III (RER With CR [ABVE-PC]) | Arm IV (RER With Less Than CR [ABVE-PC, IFRT]) | Arm V (RER With PD) | Arm VI (SER [DECA, ABVE-PC, IFRT]) | Arm VII (SER [ABVE-PC, IFRT])
Started | 52 | 381 | 382 | 571 | 42 | 153 | 153
Completed | 7 | 292 | 301 | 457 | 6 | 101 | 102
Not Completed | 45 | 89 | 81 | 114 | 36 | 52 | 51
Not completed — Death | 1 | 3 | 0 | 3 | 0 | 1 | 2
Not completed — Lack of Efficacy | 2 | 46 | 60 | 78 | 11 | 30 | 38
Not completed — Lost to Follow-up | 2 | 9 | 13 | 13 | 1 | 3 | 1
Not completed — Physician Decision | 12 | 1 | 0 | 5 | 4 | 2 | 1
Not completed — Protocol Violation | 3 | 2 | 2 | 1 | 2 | 1 | 3
Not completed — Withdrawal by Subject | 9 | 27 | 6 | 14 | 11 | 8 | 3
Not completed — Ineligible | 14 | 1 | 0 | 0 | 6 | 0 | 1
Not completed — Randomization error | 1 | 0 | 0 | 0 | 1 | 7 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Patients Off-therapy Before Callback-Induction Only) | Arm II (RER With CR [ABVE-PC, IFRT]) | Arm III (RER With CR [ABVE-PC]) | Arm IV (RER With Less Than CR [ABVE-PC, IFRT]) | Arm V (RER With PD) | Arm VI (SER [DECA, ABVE-PC, IFRT]) | Arm VII (SER [ABVE-PC, IFRT]) | Total
Number analyzed (Participants) | 52 | 381 | 382 | 571 | 42 | 153 | 153 | 1734
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 46 | 363 | 369 | 540 | 40 | 143 | 148 | 1649
  Between 18 and 65 years | 6 | 18 | 13 | 31 | 2 | 10 | 5 | 85
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: Years] | 16 [5 to 20] | 14 [2 to 21] | 14 [3 to 21] | 15 [1 to 21] | 15 [5 to 19] | 15 [5 to 21] | 15 [5 to 21] | 15 [1 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 177 | 155 | 288 | 16 | 81 | 77 | 815
  Male | 31 | 204 | 227 | 283 | 26 | 72 | 76 | 919
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 71 | 67 | 74 | 4 | 22 | 14 | 259
  Not Hispanic or Latino | 44 | 293 | 306 | 487 | 34 | 127 | 134 | 1425
  Unknown or Not Reported | 1 | 17 | 9 | 10 | 4 | 4 | 5 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 4
  Asian | 1 | 15 | 12 | 11 | 1 | 4 | 6 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 6
  Black or African American | 5 | 45 | 43 | 67 | 6 | 14 | 14 | 194
  White | 41 | 290 | 297 | 444 | 30 | 122 | 124 | 1348
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 31 | 27 | 45 | 4 | 12 | 8 | 132
Region of Enrollment [Number; unit: participants]
  New Zealand | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 4
  Canada | 8 | 30 | 45 | 51 | 1 | 20 | 20 | 175
  United States | 41 | 333 | 312 | 491 | 39 | 125 | 128 | 1469
  Israel | 0 | 3 | 1 | 1 | 0 | 1 | 0 | 6
  Australia | 0 | 8 | 13 | 12 | 0 | 3 | 4 | 40
  Switzerland | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Kuwait | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  France | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Netherlands | 0 | 2 | 9 | 7 | 1 | 3 | 0 | 22
  Puerto Rico | 1 | 4 | 2 | 4 | 0 | 1 | 1 | 13
  Bermuda | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  French Polynesia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival
Description: Probability of event-Free survival which is defined as the time from study entry to treatment failure (disease progression, disease recurrence, biopsy positive residual after completion of all protocol therapy), occurrence of a second malignant neoplasm, or death from any cause. Patients without report of such events where censored at last contact.
Time Frame: 5 years
Population: Eligible participants are analyzed and ineligible participants (n=22) are excluded from Arms I (n=14), II (n=1), III (n=0), IV (n=6), V (n=0), VI (n=1), and VII (n=0).
Measure: Number (95% Confidence Interval); unit: Probability of survival
Groups:
- Arm I (Patients Off-therapy Before Callback-Induction Only): All patients-off therapy before callback-Induction only
- Arm II (RER With CR [ABVE-PC, IFRT]): RER with Complete Response - IFRT (Standard Arm)
- Arm III (RER With CR [ABVE-PC]): RER with Complete Response - no IFRT (Reduced Therapy Arm)
- Arm IV (RER With Less Than CR [ABVE-PC, IFRT]): RER with less than Complete Response - IFRT
- Arm V (RER With PD): RER with Progressive Disease - Off Therapy
- Arm VI (SER [DECA, ABVE-PC, IFRT]): SER - randomized to DECAX2 + ABVE-PCX2 + IFRT
- Arm VII (SER [ABVE-PC, IFRT]): SER - randomized to ABVE-PCX2 + IFRT
Arm/Group | Arm I (Patients Off-therapy Before Callback-Induction Only) | Arm II (RER With CR [ABVE-PC, IFRT]) | Arm III (RER With CR [ABVE-PC]) | Arm IV (RER With Less Than CR [ABVE-PC, IFRT]) | Arm V (RER With PD) | Arm VI (SER [DECA, ABVE-PC, IFRT]) | Arm VII (SER [ABVE-PC, IFRT])
Number analyzed (Participants) | 38 | 380 | 382 | 571 | 36 | 153 | 152
Probability of survival | 0.89 [0.69 to 0.96] | 0.87 [0.83 to 0.90] | 0.84 [0.80 to 0.87] | 0.87 [0.83 to 0.89] | 0.70 [0.51 to 0.82] | 0.79 [0.71 to 0.85] | 0.74 [0.66 to 0.80]

2. Secondary Outcome: Disease Response Assessed by Modified RECIST Criteria
Description: Number of participants with complete response and very good partial response at the end of protocol therapy.
Time Frame: Protocol therapy: the overall duration of which is: (n=1527) an average of 137.1 days, median 133.0 days, interquartile range: 101.0, 164.0 days.
Population: as for outcome 1
Measure: Number; unit: Number of participants
Groups:
- Arm III (RER With CR [ABVE-PC]): RER with Complete Response - no IFRT ( Reduced Therapy Arm)
Arm/Group | Arm I (Patients Off-therapy Before Callback-Induction Only) | Arm II (RER With CR [ABVE-PC, IFRT]) | Arm III (RER With CR [ABVE-PC]) | Arm IV (RER With Less Than CR [ABVE-PC, IFRT]) | Arm V (RER With PD) | Arm VI (SER [DECA, ABVE-PC, IFRT]) | Arm VII (SER [ABVE-PC, IFRT])
Number analyzed (Participants) | 38 | 380 | 382 | 571 | 36 | 153 | 152
Number of participants | 5 | 370 | 380 | 538 | 29 | 105 | 100

3. Secondary Outcome: Grade 3 or 4 Non-hematologic Toxicity
Description: Occurrence of any grade 4 non-hematologic toxicity or grade 3 non-hematologic toxicity which doesn't respond to treatment within 7 days despite recommended therapy modification, or toxic death, which is any death primarily attributable to treatment. Grade 3 is defined to be severe or medically significant but not immediate life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 refers to toxicities with life-threatening consequences; urgent intervention indicated.
Time Frame: Protocol therapy: the overall duration of which is: (n=1684) an average of 137.3 days, median 133.0 days, interquartile range: 101.0, 164.0 days.
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Arm I (Patients Off-therapy Before Callback-Induction Only) | Arm II (RER With CR [ABVE-PC, IFRT]) | Arm III (RER With CR [ABVE-PC]) | Arm IV (RER With Less Than CR [ABVE-PC, IFRT]) | Arm V (RER With PD) | Arm VI (SER [DECA, ABVE-PC, IFRT]) | Arm VII (SER [ABVE-PC, IFRT])
Number analyzed (Participants) | 38 | 380 | 382 | 571 | 36 | 153 | 152
Number of participants | 10 | 153 | 130 | 216 | 11 | 62 | 45

4. Secondary Outcome: Overall Survival
Description: Probability of overall survival which is defined as the time from study entry to death from any cause. Patients alive where censored at last contact.
Time Frame: 5 years
Population: Arm V (RER with PD), has been excluded as there were no deaths observed by the Time Frame of 5 years. Eligible participants are analyzed and ineligible participants (n=22) are excluded from Arms I (n=14), II (n=1), III (n=0), IV (n=6), V (n=0), VI (n=1), and VII (n=0).
Measure: Number (95% Confidence Interval); unit: Probability of survival
Arm/Group | Arm I (Patients Off-therapy Before Callback-Induction Only) | Arm II (RER With CR [ABVE-PC, IFRT]) | Arm III (RER With CR [ABVE-PC]) | Arm IV (RER With Less Than CR [ABVE-PC, IFRT]) | Arm VI (SER [DECA, ABVE-PC, IFRT]) | Arm VII (SER [ABVE-PC, IFRT])
Number analyzed (Participants) | 38 | 380 | 382 | 571 | 153 | 152
Probability of survival | 0.93 [0.74 to 0.98] | 0.98 [0.96 to 0.99] | 0.98 [0.96 to 0.99] | 0.98 [0.96 to 0.99] | 0.96 [0.91 to 0.98] | 0.93 [0.87 to 0.96]

ADVERSE EVENTS:
Description: Serious AE:
  Eligible participants are analyzed and ineligible participants (n=22) are excluded from Arms I (n=14), II (n=1), III (n=0), IV (n=6), V (n=0), VI (n=1), and VII (n=0).
  Other AE:
  Eligible participants are analyzed and ineligible participants (n=22) are excluded from Arms I (n=14), II (n=1), III (n=0), IV (n=6), V (n=0), VI (n=1), and VII (n=0).
Arm/Group | Arm I (Patients Off-therapy Before Callback-Induction Only) | Arm II (RER With CR [ABVE-PC, IFRT]) | Arm III (RER With CR [ABVE-PC]) | Arm IV (RER With Less Than CR [ABVE-PC, IFRT]) | Arm V (RER With PD) | Arm VI (SER [DECA, ABVE-PC, IFRT]) | Arm VII (SER [ABVE-PC, IFRT])
Serious Adverse Events (participants affected / at risk) | 1/38 | 2/380 | 1/382 | 5/571 | 1/36 | 2/153 | 1/152
Other Adverse Events (participants affected / at risk) | 23/38 | 341/380 | 334/382 | 497/571 | 26/36 | 135/153 | 133/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Patients Off-therapy Before Callback-Induction Only) (N=38) | Arm II (RER With CR [ABVE-PC, IFRT]) (N=380) | Arm III (RER With CR [ABVE-PC]) (N=382) | Arm IV (RER With Less Than CR [ABVE-PC, IFRT]) (N=571) | Arm V (RER With PD) (N=36) | Arm VI (SER [DECA, ABVE-PC, IFRT]) (N=153) | Arm VII (SER [ABVE-PC, IFRT]) (N=152)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Blood antidiuretic hormone abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Patients Off-therapy Before Callback-Induction Only) (N=38) | Arm II (RER With CR [ABVE-PC, IFRT]) (N=380) | Arm III (RER With CR [ABVE-PC]) (N=382) | Arm IV (RER With Less Than CR [ABVE-PC, IFRT]) (N=571) | Arm V (RER With PD) (N=36) | Arm VI (SER [DECA, ABVE-PC, IFRT]) (N=153) | Arm VII (SER [ABVE-PC, IFRT]) (N=152)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 196 (196) | 162 (162) | 245 (245) | 12 (12) | 85 (85) | 63 (63)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 50 (50) | 35 (35) | 57 (57) | 0 (0) | 31 (31) | 20 (20)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 111 (111) | 99 (99) | 128 (128) | 3 (3) | 45 (45) | 31 (31)
Cardiac disorders - Other, specify (Cardiac disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4) | 6 (6) | 12 (12) | 0 (0) | 1 (1) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 9 (9) | 0 (0) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 20 (20) | 9 (9) | 25 (25) | 1 (1) | 10 (10) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 6 (6) | 5 (5) | 21 (21) | 0 (0) | 6 (6) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 3 (3) | 4 (4) | 3 (3) | 7 (7) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 6 (6) | 9 (9) | 19 (19) | 0 (0) | 9 (9) | 3 (3)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 4 (4) | 4 (4) | 13 (13) | 0 (0) | 2 (2) | 0 (0)
Anaphylaxis (Immune system disorders) | 1 (1) | 14 (14) | 8 (8) | 20 (20) | 1 (1) | 4 (4) | 6 (6)
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 3 (3) | 14 (14) | 13 (13) | 17 (17) | 1 (1) | 3 (3) | 4 (4)
Infections and infestations - Other, specify (Infections and infestations) | 4 (4) | 71 (71) | 61 (61) | 79 (79) | 6 (6) | 26 (26) | 16 (16)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood antidiuretic hormone abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Carbon monoxide diffusing capacity decreased (Investigations) | 2 (2) | 11 (11) | 3 (3) | 11 (11) | 0 (0) | 3 (3) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Forced expiratory volume decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 14 (14) | 19 (19) | 53 (53) | 1 (1) | 24 (24) | 17 (17)
Neutrophil count decreased (Investigations) | 17 (17) | 319 (319) | 307 (307) | 449 (449) | 20 (20) | 126 (126) | 116 (116)
Platelet count decreased (Investigations) | 3 (3) | 152 (152) | 119 (119) | 167 (167) | 5 (5) | 98 (98) | 55 (55)
Serum amylase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 5 (5) | 71 (71) | 69 (69) | 126 (126) | 1 (1) | 50 (50) | 31 (31)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 10 (10) | 9 (9) | 0 (0) | 2 (2) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 7 (7) | 5 (5) | 4 (4) | 1 (1) | 8 (8) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 12 (12) | 7 (7) | 17 (17) | 0 (0) | 5 (5) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 7 (7) | 4 (4) | 9 (9) | 0 (0) | 2 (2) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2) | 5 (5) | 0 (0) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 7 (7) | 0 (0) | 0 (0) | 4 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 4 (4) | 3 (3) | 6 (6) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 7 (7) | 3 (3) | 6 (6) | 0 (0) | 1 (1) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 8 (8) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 5 (5) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Pyramidal tract syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 5 (5) | 5 (5) | 7 (7) | 0 (0) | 2 (2) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3) | 5 (5) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 11 (11) | 8 (8) | 13 (13) | 0 (0) | 2 (2) | 2 (2)
Thromboembolic event (Vascular disorders) | 0 (0) | 7 (7) | 2 (2) | 14 (14) | 0 (0) | 3 (3) | 3 (3)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior approval.